CLINICAL TRIAL: NCT05019768
Title: Topo-pachimetric Accelerated Epi-On Cross-linking Compared to Dresden Protocol Using Riboflavin With Vitamin E TPGS: Results of a 2-year Randomized Study
Brief Title: Topo-pachimetric Accelerated Epi-On Cross-linking Compared to Dresden Protocol Using Riboflavin With Vitamin E TPGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciro Caruso (Other)
Responsible Party: Sponsor-Investigator, Ciro Caruso, MD, Head of Corneal Transplant Center, Corneal Transplant Center, Pellegrini Hospital
Organization: Corneal Transplant Center, Pellegrini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 127
Record Dates: First submitted 2021-08-10; First posted 2021-08-25 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sCXL (Active Comparator): Standard protocol of Dresden Riboflavin-VEPTGS solution applied every 2 mins during UV UVA fluence of 3mW/cm2 UVA Irradiation time 30 minutes
  Interventions: Other: Standard CXL
- aCFXL (Experimental): Accelerated custom fast CXL protocol. The protocol has been developed on a published mathematical model that takes into consideration objective variables such as the equation governing the UVA-induced riboflavin con-sumption rate and the corneal thickness at its thinnest point.
  Riboflavin-VEPTGS solution: Epithelial lavage before UV UVA fluence of 1.8 ±0.9 mW/cm2 UVA Irradiation time 10 ± 1.5 minutes
  Interventions: Other: accelerated custom-fast CXL

INTERVENTIONS:
Other: accelerated custom-fast CXL — The accelerated custom fast CXL (aCFXL) has been developed on a published mathematical model that takes into consideration objective variables such as the equation governing the UVA-induced riboflavin consumption rate and the corneal thickness at its thinnest point. By knowing both values, the mathematical model allows to objectively calculate both the exact UVA irradiation value (intensity), expressed in mW/cm2, and the irradiation time
  Arms: aCFXL
Other: Standard CXL — The standard CXL procedure has been carried on following the Dresden protocol
  Arms: sCXL

SUMMARY:
In the present study the investigators compare the clinical outcome corneal cross linking with either the stand-ard Dresden (sCXL) or the accelerated custom-fast (aCFXL) ultraviolet A irradiation protocol using riboflavin-D-α-Tocopheryl polyethyleneglycol1000 succinate for progressive keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* documented progressive keratoconus
* changes in uncorrected distance visual acuity (UDVA) above 1.00 D
* Corrected distance visual acuity (BCVA) above 1.00 D
* spherical equivalent greater than 0.50 D

Exclusion Criteria:

* Corneal pachymetry of less than 400 µm
* less than 2000 cells/cm2,
* corneal scarring,
* nystagmus or any motility disorder that prevented a fixed gaze during the examination
* Current contact lens use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Topographical parameters | 2 years
  Maximum keratometry: diopters Mean keratometry: diopters Minimum corneal tickness: diopters

SECONDARY OUTCOMES:
Refractive parameters | 2 years
  Corrected distance acuity (BCVA): Logarithm of the Minimum Angle of Resolution (logMAR)
Refractive parameters | 2 years
  Spherical equi-valent: diopters Refractive cylinder magnitude: diopters
Biomechanical parameters | 2 years
  Corneal hysteresis: mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Pellegrini Hospital, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caruso C, Ostacolo C, Epstein RL, Barbaro G, Troisi S, Capobianco D. Transepithelial Corneal Cross-Linking With Vitamin E-Enhanced Riboflavin Solution and Abbreviated, Low-Dose UV-A: 24-Month Clinical Outcomes. Cornea. 2016 Feb;35(2):145-50. doi: 10.1097/ICO.0000000000000699. PMID 26606293
- [Background] Caruso C, Epstein RL, Ostacolo C, Pacente L, Troisi S, Barbaro G. Customized Corneal Cross-Linking-A Mathematical Model. Cornea. 2017 May;36(5):600-604. doi: 10.1097/ICO.0000000000001160. PMID 28257382